CLINICAL TRIAL: NCT05814926
Title: Pharmacokinetics, Safety and Tolerability of GP681 Single Oral Dose in Male and Female Patients With Different Degrees of Hepatic Impairment (Child-Pugh Classification A and B) as Compared With GP681 Administration to Male and Female Healthy Subjects
Brief Title: GP681 in Volunteers With Hepatic Impairment Compared With Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP681-202203
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers; Hepatic Impairment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Control (Experimental): Each healthy participant will receive a single dose of GP681
  Interventions: Drug: GP681
- Mild, Child-Pugh A (Experimental): Each participant with Child-Pugh A will receive a single dose of GP681
  Interventions: Drug: GP681
- Moderate; Child-Pugh B (Experimental): Each participant with Child-Pugh B will receive a single dose of GP681
  Interventions: Drug: GP681

INTERVENTIONS:
Drug: GP681 — GP681, tablet, oral

SUMMARY:
The primary objective of this study is to test whether mild (Child-Pugh A, score 5-6) and moderate (Child-Pugh B, score 7-9) hepatic impairment affects pharmacokinetics, safety and tolerability of GP681, compared with a control group with normal hepatic function following oral administration of GP681 as single dose.

DETAILED DESCRIPTION:
This is a multicenter, open-label, parallel group, single-dose study to compare pharmacokinetics of GP681 after a single 40mg oral dose in eight healthy subjects and eight mild or eight moderate hepatic impairment subjects. Subjects with hepatic impairment will be enrolled into either mild (Child-Pugh A, score 5-6) or moderate (Child-Pugh B, score 7-9) hepatic impairment groups. The healthy subjects will match with impaired hepatic function patients on ethnic group, sex(+/- 1 subject), age (+/- 10 years) and weight (+/- 25%).

Participants will be admitted into the Clinical Research Units(CRU) on Day-1. On the morning of Day 1, subjects will receive a single 40 mg oral dose of GP681 following an overnight fast (i.e., at least 10 hours). Participants will be confined to the CRU until discharge on Day 12, with PK blood sample draws for measurement of GP681 and its main metabolites being taken throughout the confinement.

Safety assessments will include physical examinations, ECGs, vital signs, standard clinical laboratory evaluations (hematology, blood chemistry, urinalysis, coagulation), AE and serious adverse event (SAE) monitoring.

All participants will have a post-study safety follow-up contact conducted approximately 12 days after administration of study treatment. The study will be considered complete once all the participants have finished the required assessments, dropped out, or been lost to follow-up before completing the required assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants，between the ages of 18 and 68 years of age (inclusive) at the time of Screening;
2. Body weight ≥50 kg for males, ≥45kg for females, and body mass index (BMI) between18-30 kg/m^2(inclusive);
3. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions.

Participants with Hepatic Impairment Only:

Participants must satisfy the criteria for primary liver disease as evidenced by a Child-Pugh A (score 5-6), B (score 7-9). Treatment-naïve participants for at least 4 weeks before screening can be entered into the study. Unless otherwise stated, participants must have been on stable doses and regimens of the concomitant medication for at least 4 weeks before screening.

Participants with Normal Hepatic Function Only:

1. Healthy participants, between the ages of 18 and 68 years of age (inclusive) at the time of Screening, matched to participants with hepatic impairment with regard to age (+/-10 years), and gender(+/-1 subject);
2. Body weight ≥50 kg for males, ≥45kg for females, and body mass index (BMI) between18-30 kg/m^2(inclusive), matched to participants with hepatic impairment with regard to body weight (+/-25% kg);
3. In good health, determined by no clinically significant findings from vital signs, physical examination, 12-lead electrocardiogram (ECG), clinical laboratory evaluations, and other safety examinations at screening, as assessed by the investigator.
4. Men must agree to use protocol-specified contraception and also to not donate sperm throughout the study and for at least 3 months after the final dose of study drug
5. Adequate hepatic function within 14 days before drug administration defined as: AST or ALT ≤ 1.5 times the upper limit of normal values, total bilirubin within normal limits.

Exclusion Criteria:

1. History of allergic conditions or allergic diseases, or a history of allergic reactions attributed to drugs. Those who cannot follow a uniform diet for special dietary requirements.
2. History of seizure，including any febrile seizure, or transient ischemic attack, or any condition that may pre-dispose to seizure (such as prior stroke, brain arteriovenous malformation, brain trauma with requiring hospitalization, and lacunar cerebral infarction).
3. Have a malignant tumor or a history of malignant tumor in the 5 years prior to screening (except for patients with non-melanoma skin cancers with no evidence of recurrence, or patients with excised cervical intraepithelial neoplasia).
4. Subjects with severe infection, trauma, gastrointestinal surgery or other major surgical operations within 4 weeks before screening;
5. Abnormal blood pressure response, or clinically significant abnormal blood pressure assessed by the investigator.
6. Having a history of clinically significant ECG abnormalities (history of tachycardia/bradycardia requiring medical therapy, II-III degree atrioventricular block, or QTcF>450ms for males，>460ms for females(corrected by Fridericia's formula), or other clinically significant abnormals assessed by the investigator.
7. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2, according to the modification of diet in renal disease equation.
8. Those who plan to undergo surgery, or intent to intent to be hospitalized during the trial.
9. A positive test for HIV antibody at screening.
10. Received any drugs that inhibit or induce the CYP450 enzyme (i.e., phenytoin, rifampin, carbamazepine, fluvoxamine, enoxacin, ticlopidine, gemfibrozil, clopidogrel, clarithromycin, itraconazole, ketoconazole, ritonavir) 4 weeks prior to screening period.
11. Received any drugs (including Chinese herbal medicine, vitamins and supplements) within 14 days or 5-half-lives (which is longer) prior to dosing;
12. Participation in another clinical trial within 3 months before dosing.
13. Those who have lost blood or donated up to 200 mL within 3 months before dosing, or those who plan to donate blood within 1 month after the end of this study.
14. Smoking more than 5 cigarettes per day within 3 months prior to screening，or who cannot stop using any tobacco products during the study period.
15. Average weekly intake of alcohol is more than 14 units alcohol (1 units ≈ 360 mL beer, or 45 mL spirits with 40% content, or 150 mL wine) within the 6 months prior to dosing, or a positive ethanol breath test at screening.
16. Substance abuse or use of soft drugs (e.g., marijuana) or use of hard drugs (e.g., cocaine, amphetamines, phenylcyclohexidine, etc.); Or screening for positive urine drug abuse (drug) tests.
17. Habitual or excessive consumption (more than 8 cups, 1cup=250mL) of grapefruit juice, tea, coffee and/or caffeinated beverages.
18. Subjects who are intolerant to venipuncture or have a history of fainting blood or acupuncture.
19. Those who have received vaccine within 1 month before screening.
20. Pregnant or lactating women, or those with positive blood pregnancy tests.
21. Male or female subjects of childbearing age agreed to take effective and safe contraception during treatment and 3 months after treatment.
22. Subjects with poor compliance, or not suitable for this study as judged by the investigator.

Participants with Hepatic Impairment Only:

1. Have received liver transplant at any time in the past.
2. Patients complicated with drug-induced liver injury.
3. Other causes of acute liver injury.
4. Patients with liver failure, or combined with hepatic encephalopathy, hepatocellular carcinoma, and esophageal and gastric variceal bleeding and other complications considered by the investigator as unsuitable for the clinical study.
5. Any history of clinically serious illness or disease or condition except for primary liver disease that the investigator believes may affect the results of the trial, including but not limited to a history of circulatory, endocrine, nervous, digestive, urinary, or hematological, immune, psychiatric, and metabolic disorders.

Participants with Normal Hepatic Function Only:

1. Any history of clinically serious illness or disease or condition except for primary liver disease that the investigator believes may affect the results of the trial, including but not limited to a history of circulatory, endocrine, nervous, digestive, urinary, or hematological, immune, psychiatric, and metabolic disorders.
2. Any history of hepatic impairment, or potential presence of liver function impairment by physical examination and laboratory examination at screening.
3. Positive result of any indicators of hepatitis B surface antigen, hepatitis C antibody within 1 week prior to screening or at screening.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of the analyte in plasma after oral administration of GP681 | Day 1 to Day12
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration after oral administration of GP681 | Day 1 to Day12
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after oral administration of GP681 | Day 1 to Day12

SECONDARY OUTCOMES:
Time to Cmax (Tmax) of the analyte in plasma | Day 1 to Day12
Terminal elimination half-life (t1/2) of the analyte in plasma | Day 1 to Day12
Apparent Clearance (CLz/F) of the analyte in plasma | Day 1 to Day12
Apparent volume of distribution (Vz/F) of the analyte in plasma | Day 1 to Day12
Number of participants with drug-related adverse events as assessed by CTCAE v5.0 | Day 1 to Day12

CONTACTS AND LOCATIONS:
Overall Officials: Haibin Yu, Principal Investigator — Beijing YouAn Hospital; Bin Xu, Principal Investigator — Beijing YouAn Hospital
Locations (1):
- Beijing You'an Hospital, Beijing Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No